CLINICAL TRIAL: NCT06160674
Title: Vowel Segmentation for Classification of Chronic Obstructive Pulmonary Disease Using Machine Learning
Status: Active, not recruiting | Type: Observational
Sponsor: Blekinge Institute of Technology (Other)
Collaborators: Excellence Center at Linköping - Lund in Information Technology (ELLIIT) (Unknown)
Responsible Party: Sponsor
Other Study IDs: BTH-6.1.1-0169-2023
Record Dates: First submitted 2023-11-28; First posted 2023-12-07 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Segmentation; Classification; COPD; Machine Learning
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD: 30 COPD participants, 16 Female and 14 Male.
  Interventions: Other: COPD
- HC: 38 HC participants, 20 Female and 18 Male.
  Interventions: Other: COPD

INTERVENTIONS:
Other: COPD — A vowel segmentation data set consisting of information from COPD and HC groups will be used to experiment with the classification performance of several Machine Learning techniques on different segments of a vowel recording.
  Other Names: HC

SUMMARY:
This work aims to evaluate whether the segmentation of vowel recordings collected from patients diagnosed with COPD and healthy control groups can increase the classification precision of machine learning techniques.

DETAILED DESCRIPTION:
Voice data and sociodemographic data on gender and age will be collected through the "VoiceDiganostic" application from the company Voice Diagnostic. Collected vowel recordings will be segmented and tested to determine whether some segments contain more information for the discrimination of COPD from healthy control groups.

Each segment will be transformed into mathematical vocal measures called voice features. A dataset consisting of voice features in conjunction with demographics and health data will be constructed for each segment which in turn will be evaluated for classification performance using several machine learning algorithms.

Descriptive statistical analysis will be held on attributes containing information on input data and gained outcomes from ML algorithms. The achieved results will be presented in the form of summary tables and graphs.

ELIGIBILITY:
Inclusion Criteria:

* being 18 years old and older.

Exclusion Criteria:

* being under 18 years old and older.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Data will be collected from participants 18 years old and older with and without COPD diagnosis will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2023-11-28 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Classification performance | 30 weeks
  Binary classification performance of the ML algorithm on each segment.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Sanmartin Berglund, MD, PhD, Principal Investigator — Blekinge Institute of Technology
Locations (1):
- Blekinge Institute of Technology, Karlskrona, Blekinge County, Sweden

IPD SHARING:
Plan to Share IPD: No
Participant data can not be shared due to the GDPR. However, the dataset created can be available upon request from the institution.

REFERENCES:
- [Derived] Idrisoglu A, Moraes ALD, Cheddad A, Anderberg P, Jakobsson A, Berglund JS. Vowel segmentation impact on machine learning classification for chronic obstructive pulmonary disease. Sci Rep. 2025 Mar 22;15(1):9930. doi: 10.1038/s41598-025-95320-3. PMID 40121302